CLINICAL TRIAL: NCT03686124
Title: Phase 1/2 Study Evaluating Genetically Modified Autologous T Cells Expressing a TCR Recognizing a Cancer/Germline Antigen as Monotherapy or in Combination With Nivolumab in Patients With Recurrent and/or Refractory Solid Tumors
Brief Title: ACTengine® IMA203/IMA203CD8 as Monotherapy or in Combination With Nivolumab in Recurrent and/or Refractory Solid Tumors
Acronym: ACTengine
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Immatics US, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IMA203-101
Record Dates: First submitted 2018-09-25; First posted 2018-09-26 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Refractory Cancer; Recurrent Cancer; Solid Tumor, Adult; Cancer
Keywords: T-cell therapy; immunotherapy; Melanoma (Skin); Melanoma, Uveal; Ovarian Carcinoma; Uterine Carcinoma; Uterine Carcinosarcoma; Immatics
MeSH Terms: conditions — Neoplasms; Recurrence; Melanoma; Uveal Melanoma; Ovarian Neoplasms | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (12):
- Dose Escalation A (closed to enrollment) (Experimental): Dose escalation of IMA203
  Interventions: Biological: IMA203 Product; Device: IMADetect®
- Extension Cohort A (Experimental): IMA203 at RP2D
  Interventions: Biological: IMA203 Product; Device: IMADetect®
- Extension Cohort B (closed to enrollment) (Experimental): IMA203 at RP2D + nivolumab
  Interventions: Biological: IMA203 Product; Drug: Nivolumab
- Extension Cohort AA (Experimental): IMA203 at final RP2D (flat dose)
  Interventions: Biological: IMA203 product- flat dose; Device: IMADetect®
- Uveal Melanoma (Experimental): IMA203 at RP2D
  Interventions: Biological: IMA203 Product; Device: IMADetect®
- Dose Escalation B (Experimental): Dose escalation of IMA203CD8
  Interventions: Biological: IMA203CD8 Product; Device: IMADetect®
- Extension Cohort C (Experimental): IMA203CD8 at dose levels confirmed to be safe
  Interventions: Biological: IMA203CD8 Product; Device: IMADetect®
- Extension Cohort D (Experimental): IMA203CD8 at dose levels confirmed to be safe; without IL-2
  Interventions: Biological: IMA203CD8 Product; Device: IMADetect®
- Ovarian (Experimental): IMA203CD8 monotherapy at dose levels confirmed to be safe
  Interventions: Biological: IMA203CD8 Product; Device: IMADetect®
- Endometrial (Experimental): IMA203CD8 monotherapy at dose levels confirmed to be safe
  Interventions: Biological: IMA203CD8 Product; Device: IMADetect®
- Head and Neck, Lung, and Triple Negative Breast Cancer (Experimental): IMA203CD8 monotherapy at dose levels confirmed to be safe
  Interventions: Biological: IMA203CD8 Product; Device: IMADetect®
- Rare Cancers (Experimental): IMA203CD8 monotherapy at dose levels confirmed to be safe
  Interventions: Biological: IMA203CD8 Product; Device: IMADetect®

INTERVENTIONS:
Biological: IMA203 Product — The cell dose will be based on viable CD3+CD8+ HLA- Dextramer+ cells per body surface area (BSA) as defined by the Mosteller formula
  Other Names: anzutresgene autoleucel; anzu-cel
  Arms: Dose Escalation A (closed to enrollment); Extension Cohort A; Extension Cohort B (closed to enrollment); Uveal Melanoma
Biological: IMA203 product- flat dose — The cell dose will be based on viable CD3+CD8+ HLA- Dextramer+ cells
  Other Names: anzutresgene autoleucel; anzu-cel
  Arms: Extension Cohort AA
Biological: IMA203CD8 Product — The cell dose will be based on viable CD3+CD8+ HLA- Dextramer+ cells per body surface area (BSA) as defined by the Mosteller formula
  Arms: Dose Escalation B; Endometrial; Extension Cohort C; Extension Cohort D; Head and Neck, Lung, and Triple Negative Breast Cancer; Ovarian; Rare Cancers
Drug: Nivolumab — Nivolumab will be given post IMA203/IMA203CD8 infusion, after hematologic recovery is achieved. Clinical supply provided by Bristol Myers Squibb.
  Other Names: Opdivo®
  Arms: Extension Cohort B (closed to enrollment)
Device: IMADetect® — IMADetect® is developed as a companion diagnostic to aid in selecting patients with relapsed and/or refractory solid cancers who might be eligible for enrollment in Immatics clinical trials.
  Arms: Dose Escalation A (closed to enrollment); Dose Escalation B; Endometrial; Extension Cohort A; Extension Cohort AA; Extension Cohort C; Extension Cohort D; Head and Neck, Lung, and Triple Negative Breast Cancer; Ovarian; Rare Cancers; Uveal Melanoma

SUMMARY:
The study's purpose is to establish the safety and tolerability of IMA203/IMA203CD8 products with or without combination with nivolumab in patients with solid tumors that express preferentially expressed antigen in melanoma (PRAME).

DETAILED DESCRIPTION:
SCREENING: Patient eligibility will be determined by protocol inclusion/exclusion criteria including HLA (human leukocyte antigen) screening and a biopsy (or collection of archival tumor tissue) for biomarker screening. If the patient is eligible, white blood cells will be taken during leukapheresis for the manufacture of IMA203 or IMA203CD8 product.

MANUFACTURING: IMA203 or IMA203CD8 products will be made from the patients' white blood cells.

TREATMENT: Lymphodepletion with cyclophosphamide and fludarabine will occur in the days before the IMA203/IMA203CD8 product infusion to improve the duration of time that IMA203/IMA203CD8 product stays in the body. The patient will be admitted to the hospital during the T-cell infusion.

After the IMA203/IMA203CD8 product infusion, if applicable, a low dose of IL-2 will be given subcutaneously until day 10.

In Extension Cohort B (IMA203) nivolumab will be administered intravenously.

Patients will be monitored closely throughout the study. The follow-up phase ends 5 years post infusion.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have recurrent/progressing and/or refractory solid tumors and must have received or not be eligible for all available indicated standard of care treatment.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* HLA-A*02:01 positive
* For patients with ovarian/fallopian tube cancer only: Patients must have confirmed diagnosis of high-grade serous or endometrioid epithelial ovarian cancer (EOC), primary peritoneal cancer, or fallopian tube cancer.
* For patients with endometrial carcinoma only: Patients must have a histologically confirmed diagnosis of recurrent or persistent endometrial carcinoma.
* Measurable disease according to RECIST 1.1
* Adequate selected organ function per protocol
* Patient's tumor must express tumor antigen by "IMADetect® RT-qPCR. Retrospective testing will be required for patients that qualify.
* Life expectancy more than 5 months
* Female patient of childbearing potential must use adequate contraception prior to study entry until 12 months after the infusion of IMA203/IMA203CD8
* Male patient must agree to use effective contraception or be abstinent while on study and for 6 months after the infusion of IMA203/IMA203CD8
* The patient must have recovered from any side effects of prior therapy to Grade 1 or lower prior to lymphodepletion.

Exclusion Criteria:

* History of other malignancies (except for adequately treated basal or squamous cell carcinoma or carcinoma in situ) within the last 3 years
* Pregnant or breastfeeding
* Serious autoimmune disease Note: At the discretion of the investigator, these patients may be included if their disease is well controlled without the use of immunosuppressive agents.
* History of cardiac conditions as per protocol
* Prior stem cell transplantation or solid organ transplantation
* Concurrent severe and/or uncontrolled medical disease that could compromise participation in the study
* History of or current immunodeficiency disease or prior treatment compromising immune function at the discretion of the treating physician
* Positive for HIV infection or with active hepatitis B virus (HBV) or active hepatitis C virus (HCV) infection.
* Patients with LDH greater than 2.0-fold ULN.
* Any condition contraindicating leukapheresis, lymphodepletion, low-dose IL-2, and/or IMA203/IMA203CD8 treatment
* Patients with active brain metastases
* Concurrent treatment in another clinical trial.
* For nivolumab treatment, patients must not have a history of severe immune-related toxicities, defined as any Grade 3 or 4 toxicities related to prior PD1/PD-L1 inhibitor therapy (e.g., atezolizumab, pembrolizumab or nivolumab etc.).

Other protocol defined inclusion/exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 375 (Estimated)
Dates: Start 2019-05-14 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2032-06 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Determine the MTD and/or recommended dose for extension for IMA203/IMA203CD8 | 28 days
  Number of patients with dose-limiting toxicities (DLTs)
Phase 1 and Phase 2: Number and grade of treatment emergent adverse events and adverse events of special interest in subjects treated. | 35 days
  Treatment emergent adverse events (TEAEs), Adverse events of special interest (AESIs) and Treatment-emergent serious adverse events (TESAEs).
Phase 1 and Phase 2: Tumor Response | 5 years
  Objective response rate (ORR) based on best overall response (BOR) of complete response (CR) and partial response (PR) centrally assessed (by a BICR1) using RECIST1.1

SECONDARY OUTCOMES:
Phase 1 and 2: Persistence of TCR engineered T-cells | up to 5 years post treatment
  Measurement of TCR-engineered T cells in peripheral blood
Phase 1 and 2: Tumor response | up to 5 years
  Overall response rate, duration of response, disease control rate and progression free survival based on Response Evaluation Criteria In Solid Tumors (RECIST) 1.1. Overall survival.
Phase 2: Patient reported quality of life | up to 5 years
  Quality of Life questionnaires (European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 and EuroQol 5-Dimension 5-Level questionnaire). Higher score indicates worsening of patient's condition.

CONTACTS AND LOCATIONS:
Overall Officials: Cedrik Britten, M.D., Study Director — Immatics US, Inc.
Locations (16):
- United States (8):
  - University of Miami Hospital and Clinics, Miami, Florida
  - University of Chicago Medical Center, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Ohio State University Wexner Medical Center Gynecologic Oncology at Mill Run, Columbus, Ohio
  - University of Pennsylvania, Perelamn Center for Advanced Medicine, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - University of Texas MD Anderson Cancer Center, Houston, Texas
- Germany (8):
  - Universitätsklinikum Heidelberg, Nationales Centrum für Tumorerkrankungen (NCT), Heidelberg, Baden-Wurttemberg
  - Klinikum rechts der Isar der Technischen Universität München, Munich, Bavaria
  - Universitätsklinikum Würzburg, Würzburg, Bavaria
  - Universitätsklinikum Bonn - Medizinische Klinik III, Bonn, North Rhine-Westphalia
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Mainz, Rhineland-Palatinate
  - Universitätsklinikum C.-G.-Carus Dresden, Dresden, Saxony
  - Charité Benjamin Franklin - Klinik für Hämatologie und Onkologie, Berlin
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg

REFERENCES:
- [Derived] Wermke M, Araujo DM, Chatterjee M, Tsimberidou AM, Holderried TAW, Jazaeri AA, Reshef R, Bokemeyer C, Alsdorf W, Wetzko K, Brossart P, Aslan K, Backert L, Bunk S, Fritsche J, Gulde S, Hengler S, Hilf N, Hossain MB, Hukelmann J, Kalra M, Krishna D, Kursunel MA, Maurer D, Mayer-Mokler A, Mendrzyk R, Mohamed A, Pozo K, Satelli A, Letizia M, Schuster H, Schoor O, Wagner C, Rammensee HG, Reinhardt C, Singh-Jasuja H, Walter S, Weinschenk T, Luke JJ, Britten CM. Autologous T cell therapy for PRAME+ advanced solid tumors in HLA-A*02+ patients: a phase 1 trial. Nat Med. 2025 Jul;31(7):2365-2374. doi: 10.1038/s41591-025-03650-6. Epub 2025 Apr 9. PMID 40205198